CLINICAL TRIAL: NCT06833164
Title: Serum ERAP1 and ERAP2 Levels in Patients With Recalcitrant Warts
Brief Title: ERAP1,2 in Recalcitrant Warts
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, karem Taha ibrahim khalil, assistant professor of dermatology, venereology and andrology, Benha University
Other Study IDs: Serum ERAP1 and 2 in warts
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: endoplasmic reticulum Aminopeptidase 1 and 2 — endoplasmic reticulum aminopeptidase1 and 2 serum levels determination via ELISA
Diagnostic Test: endoplasmic reticulum aminopeptidase 1 and 2 serum levels determination via ELISA — endoplasmic reticulum aminopeptidase 1 and 2 serum levels determination via ELISA
  Other Names: SEUM ERAP1 MEASUREMENT USING ELISA; SERUM ERAP2MEASUREMENT USING ELISA

SUMMARY:
The exact mechanisms underlying the contribution of cellular immunity in the eradication of human papillomavirus (HPV) infections remain obscure. Individuals who have treatment-resistant warts frequently have immune deficiencies. Amino-peptidases (ERAP1, ERAP2) of endoplasmic reticulum are essential for production of antigenic epitopes that attach to the Major Histocompatibility Complex (MHC) class I and activate T-lymphocytes or natural killer (NK) cells. Aim: To assess ERAP1 and ERAP2 serum concentrations in patients with resistant warts.

ELIGIBILITY:
Inclusion Criteria:

• Patients who had a history of incomplete clearance or recurrence following two or more electrocautery sessions and four or more cryocautery treatments and intralesional bleomycin.

Exclusion Criteria:

* Patients with genital warts
* Patients on systemic steroids or other immunosuppressive treatments
* Immunocompromised individuals
* Patients suffering from chronic systemic diseases
* Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred individuals were separated into two groups. Group (I) patients with resistant warts (n=100), and group (II) age- and sex-matched subjects with history of treated warts with no recurrence (n=100). They were recruited from the Dermatology Outpatient Clinic at Benha University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
SERUM LEVELS OF endoplasmic reticulum aminopeptidase 1 and 2 | ONE YEAR
  using specific Commercial human ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Y. Abdallah, MD, Study Chair — Professor of Dermatology, Venereology and Andrology, Faculty of Medicine, Benha University; Nehad A.Fouad, MD, Study Director — Professor of Microbiology and Immunology, Faculty of Medicine, Benha University; Ola S Ebrahim, MBBCh, Principal Investigator — Benha University
Locations (1):
- faculty of medicine Benha University, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided